CLINICAL TRIAL: NCT03747523
Title: Study of the Effect of Ergocalciferol on Plasma and Urinary Mucin-1 Levels in Healthy Individuals and Individuals With Autosomal Dominant Tubulo-Interstitial Kidney Disease Due to MUC1 Mutations (ADTKD-MUC1)
Brief Title: Pilot Study: The Effect of Ergocalciferol on Plasma Mucin-1 Levels
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00054784
Record Dates: First submitted 2018-11-16; First posted 2018-11-20 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-01

CONDITIONS: Ergocalciferol
Keywords: Vitamin D Deficiency; Drisdol; Rickets; Plasma; Healthy Subjects; Autosomal Dominant Tubulo Interstitial Kidney Disease
MeSH Terms: conditions — Vitamin D Deficiency; Rickets | interventions — Ergocalciferols; Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Healthy Group (Experimental): 40 Healthy individuals will receive a single dose of ergocalciferol (200,000 units)
  Interventions: Drug: Ergocalciferol
- ADTKD-MUC1 Group (Experimental): 40 individuals with ADTKD-MUC1 (Autosomal Dominant Tubulo-Interstitial Kidney Disease- a rare disease caused by mutation in MUC1) will receive a single dose of ergocalciferol (200,000 units)
  Interventions: Drug: Ergocalciferol

INTERVENTIONS:
Drug: Ergocalciferol — Investigational drug will be administered to eligible participants in a single dose of 200,000 USP units vitamin D
  Other Names: Drisdol; Calciferol; Calcidol; Vitamin D2

SUMMARY:
To determine if a one-time oral administration of ergocalciferol results in a decline in plasma mucin-1 levels in healthy individuals and individuals with ADTKD-MUC1.

DETAILED DESCRIPTION:
This is a pilot, open-labelled, to determine if oral administration of a single dose of ergocalciferol lowers plasma mucin-1 levels. The study population will include 40 healthy individuals and 40 individuals with ADTKD-MUC1.

The study consists of an initial screening, signing of consent of interested individuals, performance of pregnancy test in women of child-bearing age and screening labs, and administration of 200,000 units of ergocalciferol on Day 0 (On Study). Laboratory studies will be performed at baseline, on Days 3, 7, and 10.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years and <65 years
* Females must be non-pregnant, non-lactating and fulfilling one of the following: a. Post menopausal defined as amenorrhea for at least 12 months following cessation of all exogenous hormonal treatments. b. Status post irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation. c.

Use of acceptable contraceptive method: IUD with spermicide, a female condom with spermicide, contraceptive sponge with spermicide, an intravaginal system(e.g., NuvaRing®), a diaphragm with spermicide, a cervical cap with spermicide, or oral, implantable, transdermal, or injectable contraceptives, sexual abstinence, or a sterile sexual partner.

* Males must agree to avoid fathering a child (or donating sperm), and therefore be either sterile or agree to use, from the time of enrollment until 45 days after end of study, one of the following approved methods of contraception: a male condom with spermicide, a sterile sexual partner, use by female sexual partner of an IUD with spermicide, a female condom with spermicide, contraceptive sponge with spermicide, an intravaginal system (e.g.,NuvaRing®), a diaphragm with spermicide, a cervical cap with spermicide, or oral, implantable, transdermal, or injectable contraceptives.
* No serious health conditions except for estimated glomerular filtration rate <30 ml/min/1.73 m2 (according to the modified MDRD formula) in participants with ADTKD- MUC1.
* Prior established genetic diagnosis of ADTKD-MUC1 in participants recruited with ADTKD-MUC1.
* Able to understand and comply with requirements of the entire study and to communicate with the study team.
* Living in close enough proximity to a local laboratory to obtain labwork for the study.
* Written informed consent using a document that has been approved by the Institutional Review Board.
* The participant has not taken ergocalciferol in the month prior to study initiation. If receiving cholecalciferol, the dose is < 1000/day and has been stopped one month prior to Day 0 (On Study).
* Participants agree NOT to take ergocalciferol or cholecalciferol (except for<500 IU that contained in a daily multi-vitamin) for six months after receiving the one-time dose of ergocalciferol.

Exclusion Criteria:

* Major systemic illness other than chronic kidney disease in individuals with ADTKD- MUC1.
* A history of granulomatous disorders (sarcoidosis, tuberculosis), hyperparathyroidism, or other disorders of calcium metabolism.
* A history of nephrolithiasis.
* A history of osteoporosis or osteopenia.
* A fracture or a fall that did not occur during exercise within the last six months.
* Intolerance or known allergic reaction to ergocalciferol.
* 25 hydroxy Vitamin D level > upper limit of normal.
* Lactating.
* Liver disease.
* Receiving glucocorticoids.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2020-01-27 (Actual)

PRIMARY OUTCOMES:
Plasma mucin-1 levels | Baseline
  Plasma mucin-1 levels will be measured in both groups. using a two-tailed T-test.
Plasma mucin-1 levels | 3 days
  Plasma mucin-1 levels will be measured in both groups. using a two-tailed T-test.

SECONDARY OUTCOMES:
Plasma mucin-1 levels | 7 days
  Plasma mucin-1 levels will be measured in will be measured in both groups.
Plasma mucin-1 levels | 10 days
  Plasma mucin-1 levels will be measured in will be measured in both groups.
Urinary mucin-1 levels in healthy controls | Baseline
  Urinary mucin-1 levels
Urinary mucin-1 levels in healthy controls | 3 days
  Urinary mucin-1 levels
Urinary mucin-1 levels in healthy controls | 7 days
  Urinary mucin-1 levels
Urinary mucin-1 levels in healthy controls | 10 days
  Urinary mucin-1 levels

CONTACTS AND LOCATIONS:
Overall Officials: Anthony J. Bleyer, MD, M.S, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kirby A, Gnirke A, Jaffe DB, Baresova V, Pochet N, Blumenstiel B, Ye C, Aird D, Stevens C, Robinson JT, Cabili MN, Gat-Viks I, Kelliher E, Daza R, DeFelice M, Hulkova H, Sovova J, Vylet'al P, Antignac C, Guttman M, Handsaker RE, Perrin D, Steelman S, Sigurdsson S, Scheinman SJ, Sougnez C, Cibulskis K, Parkin M, Green T, Rossin E, Zody MC, Xavier RJ, Pollak MR, Alper SL, Lindblad-Toh K, Gabriel S, Hart PS, Regev A, Nusbaum C, Kmoch S, Bleyer AJ, Lander ES, Daly MJ. Mutations causing medullary cystic kidney disease type 1 lie in a large VNTR in MUC1 missed by massively parallel sequencing. Nat Genet. 2013 Mar;45(3):299-303. doi: 10.1038/ng.2543. Epub 2013 Feb 10. PMID 23396133
- [Background] Bleyer AJ, Kmoch S: Autosomal Dominant Tubulointerstitial Kidney Disease, MUC1-Related. 1993
- [Background] Bleyer AJ, Kmoch S, Antignac C, Robins V, Kidd K, Kelsoe JR, Hladik G, Klemmer P, Knohl SJ, Scheinman SJ, Vo N, Santi A, Harris A, Canaday O, Weller N, Hulick PJ, Vogel K, Rahbari-Oskoui FF, Tuazon J, Deltas C, Somers D, Megarbane A, Kimmel PL, Sperati CJ, Orr-Urtreger A, Ben-Shachar S, Waugh DA, McGinn S, Bleyer AJ Jr, Hodanova K, Vylet'al P, Zivna M, Hart TC, Hart PS. Variable clinical presentation of an MUC1 mutation causing medullary cystic kidney disease type 1. Clin J Am Soc Nephrol. 2014 Mar;9(3):527-35. doi: 10.2215/CJN.06380613. Epub 2014 Feb 7. PMID 24509297
- [Background] Apostolopoulos V, Stojanovska L, Gargosky SE. MUC1 (CD227): a multi-tasked molecule. Cell Mol Life Sci. 2015 Dec;72(23):4475-500. doi: 10.1007/s00018-015-2014-z. Epub 2015 Aug 21. PMID 26294353
- [Background] Horimasu Y, Hattori N, Ishikawa N, Kawase S, Tanaka S, Yoshioka K, Yokoyama A, Kohno N, Bonella F, Guzman J, Ohshimo S, Costabel U. Different MUC1 gene polymorphisms in German and Japanese ethnicities affect serum KL-6 levels. Respir Med. 2012 Dec;106(12):1756-64. doi: 10.1016/j.rmed.2012.09.001. Epub 2012 Sep 18. PMID 22995277
- [Background] Janssen R, Kruit A, Grutters JC, Ruven HJ, Gerritsen WB, van den Bosch JM. The mucin-1 568 adenosine to guanine polymorphism influences serum Krebs von den Lungen-6 levels. Am J Respir Cell Mol Biol. 2006 Apr;34(4):496-9. doi: 10.1165/rcmb.2005-0151OC. Epub 2005 Dec 15. PMID 16357367
- [Background] Ligtenberg MJ, Gennissen AM, Vos HL, Hilkens J. A single nucleotide polymorphism in an exon dictates allele dependent differential splicing of episialin mRNA. Nucleic Acids Res. 1991 Jan 25;19(2):297-301. doi: 10.1093/nar/19.2.297. PMID 2014168
- [Background] Zivna M, Kidd K, Pristoupilova A, Baresova V, DeFelice M, Blumenstiel B, Harden M, Conlon P, Lavin P, Connaughton DM, Hartmannova H, Hodanova K, Stranecky V, Vrbacka A, Vyletal P, Zivny J, Votruba M, Sovova J, Hulkova H, Robins V, Perry R, Wenzel A, Beck BB, Seeman T, Viklicky O, Rajnochova-Bloudickova S, Papagregoriou G, Deltas CC, Alper SL, Greka A, Bleyer AJ, Kmoch S. Noninvasive Immunohistochemical Diagnosis and Novel MUC1 Mutations Causing Autosomal Dominant Tubulointerstitial Kidney Disease. J Am Soc Nephrol. 2018 Sep;29(9):2418-2431. doi: 10.1681/ASN.2018020180. Epub 2018 Jul 2. PMID 29967284
- [Background] Spicer AP, Rowse GJ, Lidner TK, Gendler SJ. Delayed mammary tumor progression in Muc-1 null mice. J Biol Chem. 1995 Dec 15;270(50):30093-101. doi: 10.1074/jbc.270.50.30093. PMID 8530414
- [Background] Corsello SM, Bittker JA, Liu Z, Gould J, McCarren P, Hirschman JE, Johnston SE, Vrcic A, Wong B, Khan M, Asiedu J, Narayan R, Mader CC, Subramanian A, Golub TR. The Drug Repurposing Hub: a next-generation drug library and information resource. Nat Med. 2017 Apr 7;23(4):405-408. doi: 10.1038/nm.4306. No abstract available. PMID 28388612
- [Background] Bonella F, Long X, Ohshimo S, Horimasu Y, Griese M, Guzman J, Kohno N, Costabel U. MUC1 gene polymorphisms are associated with serum KL-6 levels and pulmonary dysfunction in pulmonary alveolar proteinosis. Orphanet J Rare Dis. 2016 Apr 23;11:48. doi: 10.1186/s13023-016-0430-2. PMID 27108412
- [Background] Estebanez N, Gomez-Acebo I, Palazuelos C, Llorca J, Dierssen-Sotos T. Vitamin D exposure and Risk of Breast Cancer: a meta-analysis. Sci Rep. 2018 Jun 13;8(1):9039. doi: 10.1038/s41598-018-27297-1. PMID 29899554
- [Background] Conley SJ, Bosco EE, Tice DA, Hollingsworth RE, Herbst R, Xiao Z. HER2 drives Mucin-like 1 to control proliferation in breast cancer cells. Oncogene. 2016 Aug 11;35(32):4225-34. doi: 10.1038/onc.2015.487. Epub 2016 Jan 4. PMID 26725324
- [Background] Nguyen B, Venet D, Azim HA Jr, Brown D, Desmedt C, Lambertini M, Majjaj S, Pruneri G, Peccatori F, Piccart M, Rothe F, Sotiriou C. Breast cancer diagnosed during pregnancy is associated with enrichment of non-silent mutations, mismatch repair deficiency signature and mucin mutations. NPJ Breast Cancer. 2018 Aug 6;4:23. doi: 10.1038/s41523-018-0077-3. eCollection 2018. PMID 30109263
- [Background] Sinn BV, von Minckwitz G, Denkert C, Eidtmann H, Darb-Esfahani S, Tesch H, Kronenwett R, Hoffmann G, Belau A, Thommsen C, Holzhausen HJ, Grasshoff ST, Baumann K, Mehta K, Dietel M, Loibl S. Evaluation of Mucin-1 protein and mRNA expression as prognostic and predictive markers after neoadjuvant chemotherapy for breast cancer. Ann Oncol. 2013 Sep;24(9):2316-24. doi: 10.1093/annonc/mdt162. Epub 2013 May 9. PMID 23661292
- [Background] Heaney RP, Armas LA, Shary JR, Bell NH, Binkley N, Hollis BW. 25-Hydroxylation of vitamin D3: relation to circulating vitamin D3 under various input conditions. Am J Clin Nutr. 2008 Jun;87(6):1738-42. doi: 10.1093/ajcn/87.6.1738. PMID 18541563
- [Background] Sanders KM, Stuart AL, Williamson EJ, Simpson JA, Kotowicz MA, Young D, Nicholson GC. Annual high-dose oral vitamin D and falls and fractures in older women: a randomized controlled trial. JAMA. 2010 May 12;303(18):1815-22. doi: 10.1001/jama.2010.594. PMID 20460620
- [Background] Yu CK, Sykes L, Sethi M, Teoh TG, Robinson S. Vitamin D deficiency and supplementation during pregnancy. Clin Endocrinol (Oxf). 2009 May;70(5):685-90. doi: 10.1111/j.1365-2265.2008.03403.x. Epub 2008 Sep 2. PMID 18771564
- [Background] Kearns MD, Alvarez JA, Tangpricha V. Large, single-dose, oral vitamin D supplementation in adult populations: a systematic review. Endocr Pract. 2014 Apr;20(4):341-51. doi: 10.4158/EP13265.RA. PMID 24246341
- [Background] Romagnoli E, Mascia ML, Cipriani C, Fassino V, Mazzei F, D'Erasmo E, Carnevale V, Scillitani A, Minisola S. Short and long-term variations in serum calciotropic hormones after a single very large dose of ergocalciferol (vitamin D2) or cholecalciferol (vitamin D3) in the elderly. J Clin Endocrinol Metab. 2008 Aug;93(8):3015-20. doi: 10.1210/jc.2008-0350. Epub 2008 May 20. PMID 18492750
- [Background] Houghton LA, Vieth R. The case against ergocalciferol (vitamin D2) as a vitamin supplement. Am J Clin Nutr. 2006 Oct;84(4):694-7. doi: 10.1093/ajcn/84.4.694. PMID 17023693
- [Background] Logan VF, Gray AR, Peddie MC, Harper MJ, Houghton LA. Long-term vitamin D3 supplementation is more effective than vitamin D2 in maintaining serum 25-hydroxyvitamin D status over the winter months. Br J Nutr. 2013 Mar 28;109(6):1082-8. doi: 10.1017/S0007114512002851. Epub 2012 Jul 11. PMID 23168298
- [Background] Armas LA, Hollis BW, Heaney RP. Vitamin D2 is much less effective than vitamin D3 in humans. J Clin Endocrinol Metab. 2004 Nov;89(11):5387-91. doi: 10.1210/jc.2004-0360. PMID 15531486
- [Background] Trang HM, Cole DE, Rubin LA, Pierratos A, Siu S, Vieth R. Evidence that vitamin D3 increases serum 25-hydroxyvitamin D more efficiently than does vitamin D2. Am J Clin Nutr. 1998 Oct;68(4):854-8. doi: 10.1093/ajcn/68.4.854. PMID 9771862
- [Background] Grossmann RE, Zughaier SM, Kumari M, Seydafkan S, Lyles RH, Liu S, Sueblinvong V, Schechter MS, Stecenko AA, Ziegler TR, Tangpricha V. Pilot study of vitamin D supplementation in adults with cystic fibrosis pulmonary exacerbation: A randomized, controlled trial. Dermatoendocrinol. 2012 Apr 1;4(2):191-7. doi: 10.4161/derm.20332. PMID 22928076
- [Background] Witham MD, Dove FJ, Dryburgh M, Sugden JA, Morris AD, Struthers AD. The effect of different doses of vitamin D(3) on markers of vascular health in patients with type 2 diabetes: a randomised controlled trial. Diabetologia. 2010 Oct;53(10):2112-9. doi: 10.1007/s00125-010-1838-1. Epub 2010 Jul 2. PMID 20596692
- [Background] Premaor MO, Scalco R, da Silva MJ, Froehlich PE, Furlanetto TW. The effect of a single dose versus a daily dose of cholecalciferol on the serum 25-hydroxycholecalciferol and parathyroid hormone levels in the elderly with secondary hyperparathyroidism living in a low-income housing unit. J Bone Miner Metab. 2008;26(6):603-8. doi: 10.1007/s00774-008-0858-0. Epub 2008 Nov 1. PMID 18979160
- [Background] Sakalli H, Arslan D, Yucel AE. The effect of oral and parenteral vitamin D supplementation in the elderly: a prospective, double-blinded, randomized, placebo-controlled study. Rheumatol Int. 2012 Aug;32(8):2279-83. doi: 10.1007/s00296-011-1943-6. Epub 2011 May 10. PMID 21556746
- [Background] Stoll D, Dudler J, Lamy O, Hans D, Krieg MA, Aubry-Rozier B. Can one or two high doses of oral vitamin D3 correct insufficiency in a non-supplemented rheumatologic population? Osteoporos Int. 2013 Feb;24(2):495-500. doi: 10.1007/s00198-012-1962-5. Epub 2012 Mar 17. PMID 22426953
- [Background] Bacon CJ, Gamble GD, Horne AM, Scott MA, Reid IR. High-dose oral vitamin D3 supplementation in the elderly. Osteoporos Int. 2009 Aug;20(8):1407-15. doi: 10.1007/s00198-008-0814-9. Epub 2008 Dec 20. PMID 19101755
- [Background] Smith H, Anderson F, Raphael H, Maslin P, Crozier S, Cooper C. Effect of annual intramuscular vitamin D on fracture risk in elderly men and women--a population-based, randomized, double-blind, placebo-controlled trial. Rheumatology (Oxford). 2007 Dec;46(12):1852-7. doi: 10.1093/rheumatology/kem240. Epub 2007 Nov 12. PMID 17998225
- [Background] Amrein K, Sourij H, Wagner G, Holl A, Pieber TR, Smolle KH, Stojakovic T, Schnedl C, Dobnig H. Short-term effects of high-dose oral vitamin D3 in critically ill vitamin D deficient patients: a randomized, double-blind, placebo-controlled pilot study. Crit Care. 2011;15(2):R104. doi: 10.1186/cc10120. Epub 2011 Mar 28. PMID 21443793
- [Background] Rossini M, Gatti D, Viapiana O, Fracassi E, Idolazzi L, Zanoni S, Adami S. Short-term effects on bone turnover markers of a single high dose of oral vitamin D(3). J Clin Endocrinol Metab. 2012 Apr;97(4):E622-6. doi: 10.1210/jc.2011-2448. Epub 2012 Feb 1. PMID 22298802
- [Background] Tellioglu A, Basaran S, Guzel R, Seydaoglu G. Efficacy and safety of high dose intramuscular or oral cholecalciferol in vitamin D deficient/insufficient elderly. Maturitas. 2012 Aug;72(4):332-8. doi: 10.1016/j.maturitas.2012.04.011. Epub 2012 May 20. PMID 22613271
- [Background] Latham NK, Anderson CS, Lee A, Bennett DA, Moseley A, Cameron ID; Fitness Collaborative Group. A randomized, controlled trial of quadriceps resistance exercise and vitamin D in frail older people: the Frailty Interventions Trial in Elderly Subjects (FITNESS). J Am Geriatr Soc. 2003 Mar;51(3):291-9. doi: 10.1046/j.1532-5415.2003.51101.x. PMID 12588571
- [Background] Leventis P, Kiely PD. The tolerability and biochemical effects of high-dose bolus vitamin D2 and D3 supplementation in patients with vitamin D insufficiency. Scand J Rheumatol. 2009 Mar-Apr;38(2):149-53. doi: 10.1080/03009740802419081. PMID 18991184
- [Background] Kearns MD, Binongo JN, Watson D, Alvarez JA, Lodin D, Ziegler TR, Tangpricha V. The effect of a single, large bolus of vitamin D in healthy adults over the winter and following year: a randomized, double-blind, placebo-controlled trial. Eur J Clin Nutr. 2015 Feb;69(2):193-7. doi: 10.1038/ejcn.2014.209. Epub 2014 Oct 1. PMID 25271011
- [Background] Jones G. Pharmacokinetics of vitamin D toxicity. Am J Clin Nutr. 2008 Aug;88(2):582S-586S. doi: 10.1093/ajcn/88.2.582S. PMID 18689406
- [Background] Lee JP, Tansey M, Jetton JG, Krasowski MD. Vitamin D Toxicity: A 16-Year Retrospective Study at an Academic Medical Center. Lab Med. 2018 Mar 21;49(2):123-129. doi: 10.1093/labmed/lmx077. PMID 29346630
- [Background] Levey AS, Bosch JP, Lewis JB, Greene T, Rogers N, Roth D. A more accurate method to estimate glomerular filtration rate from serum creatinine: a new prediction equation. Modification of Diet in Renal Disease Study Group. Ann Intern Med. 1999 Mar 16;130(6):461-70. doi: 10.7326/0003-4819-130-6-199903160-00002. PMID 10075613

DOCUMENTS (1):
  • Informed Consent Form (2019-12-12): https://cdn.clinicaltrials.gov/large-docs/23/NCT03747523/ICF_000.pdf